CLINICAL TRIAL: NCT06496152
Title: Knowledge, Attitude, and Perceptions Towards Artificial Intelligence Among Dental Students of Faculty of Dentistry, Tanta University, Egypt
Brief Title: Knowledge, Attitude, and Perceptions Towards Artificial Intelligence Among Dental Students
Status: Not yet recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Alshimaa Ibrahim Abd El Aziz Elsandoby, Assistant Lecturer of Oral health and Preventive Dentistry, Faculty of Dentistry, Tanta University, Tanta University
Other Study IDs: artificial intelligence
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Artificial Intelligence
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional

INTERVENTIONS:
Other: questionnaire — online form used to collect all information used in questionnaire

SUMMARY:
The aim of this study will be to assess knowledge, attitudes, and perceptions towards Artificial intelligence among dental students of Faculty of Dentistry, Tanta University

DETAILED DESCRIPTION:
A cross-sectional study will be adopted using an online-based questionnaire that will be sent to dental students in the Faculty of Dentistry, Tanta University. A questionnaire will be adopted from an existing similar pre validated study. The link of the survey will be created using Microsoft form and will be disseminated through various open social media groups of dental students.

ELIGIBILITY:
Inclusion Criteria:

* all dental students of Faculty of Dentistry, Tanta University

Exclusion Criteria:

* The postgraduate students

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A cross-sectional study will be adopted using an online-based questionnaire that will be sent to dental students in the Faculty of Dentistry, Tanta University. The link of the survey will be created using Microsoft form and will be disseminated through various open social media groups of dental students
Sampling Method: Non-Probability Sample
Enrollment: 371 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-02 (Estimated)

PRIMARY OUTCOMES:
The online form by questionnaire | Two months
  Knowledge, Attitude, and Perceptions Towards Artificial Intelligence Among Dental Students

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aldowah O, Almakrami A, Alghuwaynim Y, Alhutaylah M, Almansour A, Alswedan A, Alshahrani F, Alqarni S, Alkasi Y. Perceptions and Knowledge of Undergraduate Dental Students about Artificial Intelligence in Dental Schools: A Cross-sectional Study. J Contemp Dent Pract. 2024 Feb 1;25(2):148-155. doi: 10.5005/jp-journals-10024-3633. PMID 38514412